CLINICAL TRIAL: NCT03917004
Title: Correlation Analysis of the Effects of Management Pressure Goals (Controlled Hypotension) and Control Volume Goals (Cardiac Output, Stroke Volume Variability, Central Venous Pressure) on Intraoperative Blood and Visual Field Quality
Brief Title: Correlation Analysis of the Effects of Management Pressure Goals and Control Volume Goals in Patients in Spinal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Liang Bing (Other)
Responsible Party: Sponsor-Investigator, Liang Bing, Associate chief physician, Guangzhou Red Cross Hospital
Organization: Guangzhou Red Cross Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-032-01
Record Dates: First submitted 2019-03-05; First posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Hypotension,Controlled
Keywords: controlled hypotension; cardiac output on; blood loss; surgical field; oxygen supply; oxygen consumption
MeSH Terms: conditions — Hypotension; Hemorrhage | interventions — Nitroglycerin; Hypotension, Controlled

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hypotension group (group H ) (Experimental): particcipants in hypotension group are received controlled hypertension in the operation.
  Interventions: Drug: Nitroglycerin
- control group (group C ) (No Intervention): participants in cotrol group are received no controlled hypertension in the operation

INTERVENTIONS:
Drug: Nitroglycerin — The starting rate of "nitroglycerin" was 0.25 μg / kg / min and the mean arterial pressure (MAP) decreased to 80% of the baseline but not less than 70%.The drug infusion rate was adjusted so that the MAP was maintained in the range to the suture, and the administration was stopped and the blood pressure was gradually returned to the pre-depressurization level.
  Other Names: Controlled Hypotension
  Arms: hypotension group (group H )

SUMMARY:
The investigators study 160 patients undergoing spinal surgery.Participants will be randomly divided into study group and control group.The study group will receive controlled hypotension by nitroglycerin and be divided into 3 groups according to CI.

DETAILED DESCRIPTION:
This study will be done in Guangzhou Red Cross Hospital .The investigators study 160 patients aged from 45 to 70 years,weight from 48 to 68kg classified as American Society of Anesthesiologists (ASAs) physical status Ⅰ-Ⅱ who will be candidate for posterior decompression of vertebral canal,discectomy and internal fixation by pediclescrew(one centrum).The investigators excluded patients with cardiovascular and cerebrovascular diseases,hepatic or renal dysfunction,and patients receiving drugs that interfere with coagulation before surgery.

Patients randomly divided into study group(group H,n=120)and control group (group C,n=40).The study group according to CI(Cardiac Index) levels of intraoperative hypotension period(mean of CI at T2,T3,T4) were divided into three groups: 1st group: CI: 1.5-2.0 L /(min•m2), 2nd group: CI: 2.0-3.0 L /(min•m2), 3rd group: CI: 3.0-4.0 L /(min•m2),and which CI < 1.5 or CI > 4.0 was eliminated the experimental group, which, in control group, CI< 2.5 or CI >4.0 was eliminated the experimental group.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 35 and 70 years
2. Patients, undergoing canal decompression, intervertebral disc extraction and pedicle screw fixation (1 vertebral body)

Exclusion Criteria:

1. History of cardiovascular function

   1. congestive heart failure [CHF]
   2. coronary artery disease [CAD]
   3. cerebrovascular insuffiency)
2. poorly controlled arterial hypertension
3. pre-existing coagulation defects
4. Patients taking anticoagulatory medication including aspirin
5. Patients taking corticosteroid therapy

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
cardiac index(CI) after the participants are taken into the operating room | during surgery
  CI(L/min/m^2)
cardiac index(CI) after the induction | during surgery
  cardiac index (CI,L/min/m^2)
cardiac index(CI) at 5 minutes after tubation | 5 minutes after tubation
  cardiac index (CI,L/min/m^2)
cardiac index(CI) at 10 minutes after tubation | 10 minutes after tubation
  cardiac index (CI,L/min/m^2).
cardiac index(CI) at 15 minutes after tubation | 15 minutes after tubation
  cardiac index (CI,L/min/m^2)
cardiac index(CI) at 30 minutes after tubation | 30 minutes after tubation
  cardiac index (CI,L/min/m^2)
cardiac index(CI) at 45 minutes after tubation | 45 minutes after tubation
  cardiac index (CI,L/min/m^2)
cardiac index(CI) at the end of surgery | at the end of surgery
  cardiac index (CI,L/min/m^2).
cardiac index(CI) at 1 minute after extubation | 1 minute after extubation
  cardiac index (CI,L/min/m^2)
cardiac index(CI) at 5 minutes after extubation | 5 minutes after extubation
  cardiac index (CI,L/min/m^2)

SECONDARY OUTCOMES:
Partial pressure of oxygen after the participants are taken into the operating room | during surgery
  Partial pressure of oxygen (PaO2,mmHg)
Arterial oxygen saturation after the participants are taken into the operating room | during surgery
  Arterial oxygen saturation (SaO2,%)
Arterial blood hemoglobin after the participants are taken into the operating room | during surgery
  Arterial blood hemoglobin (Hb,g/L)
Arterial blood lactate after the participants are taken into the operating room | during surgery
  Arterial blood lactate (Lac,mmol/L)
Partial pressure central venous oxygen after the participants are taken into the operating room | during surgery
  Partial pressure central venous oxygen(PvO2,mmHg)
Central venous blood oxygen saturation after the participants are taken into the operating room | during surgery
  Central venous blood oxygen saturation(ScvO2,%)
Oxygen supply index after the participants are taken into the operating room | during surgery
  Oxygen supply index (DO2I,ml/min/m^2)
Oxygen consumption index after the participants are taken into the operating room | during surgery
  Oxygen consumption index (VO2I,ml/min/m^2)
Partial pressure of oxygen after the induction | during surgery
  Partial pressure of oxygen (PaO2,mmHg)
Arterial oxygen saturation after the induction | during surgery
  Arterial oxygen saturation (SaO2,%)
Arterial blood hemoglobin after the induction | during surgery
  Arterial blood hemoglobin (Hb,g/L)
Arterial blood lactate after the induction | during surgery
  Arterial blood lactate (Lac,mmol/L)
Partial pressure central venous oxygen after the induction | during surgery
  Partial pressure central venous oxygen(PvO2,mmHg)
Central venous blood oxygen saturation after the induction | during surgery
  Central venous blood oxygen saturation(ScvO2,%)
Oxygen supply index after the induction | during surgery
  Oxygen supply index (DO2I,ml/min/m^2)
Oxygen consumption index after the induction | during surgery
  Oxygen consumption index (VO2I,ml/min/m^2)
Partial pressure of oxygen at 5 minutes after tubation | 5 minutes after tubation
  Partial pressure of oxygen (PaO2,mmHg)
Arterial oxygen saturation at 5 minutes after tubation | 5 minutes after tubation
  Arterial oxygen saturation (SaO2,%)
Arterial blood hemoglobin at 5 minutes after tubation | 5 minutes after tubation
  Arterial blood hemoglobin (Hb,g/L)
Arterial blood lactate at 5 minutes after tubation | 5 minutes after tubation
  Arterial blood lactate (Lac,mmol/L)
Partial pressure central venous oxygen at 5 minutes after tubation | 5 minutes after tubation
  Partial pressure central venous oxygen(PvO2,mmHg)
Central venous blood oxygen saturation at 5 minutes after tubation | 5 minutes after tubation
  Central venous blood oxygen saturation(ScvO2,%)
Oxygen supply index at 5 minutes after tubation | 5 minutes after tubation
  Oxygen supply index (DO2I,ml/min/m^2)
Oxygen consumption index at 5 minutes after tubation | 5 minutes after tubation
  Oxygen consumption index (VO2I,ml/min/m^2)
Partial pressure of oxygen at 10 minutes after tubation | 10 minutes after tubation
  Partial pressure of oxygen (PaO2,mmHg)
Arterial oxygen saturation at 10 minutes after tubation | 10 minutes after tubation
  Arterial oxygen saturation (SaO2,%)
Arterial blood hemoglobin at 10 minutes after tubation | 10 minutes after tubation
  Arterial blood hemoglobin (Hb,g/L)
Arterial blood lactate at 10 minutes after tubation | 10 minutes after tubation
  Arterial blood lactate (Lac,mmol/L)
Partial pressure central venous oxygen at 10 minutes after tubation | 10 minutes after tubation
  Partial pressure central venous oxygen(PvO2,mmHg)
Central venous blood oxygen saturation at 10 minutes after tubation | 10 minutes after tubation
  Central venous blood oxygen saturation(ScvO2,%)
Oxygen supply index at 10 minutes after tubation | 10 minutes after tubation
  Oxygen supply index (DO2I,ml/min/m^2)
Oxygen consumption index at 10 minutes after tubation | 10 minutes after tubation
  Oxygen consumption index (VO2I,ml/min/m^2)
Partial pressure of oxygen at 15 minutes after tubation | 15 minutes after tubation
  Partial pressure of oxygen (PaO2,mmHg)
Arterial oxygen saturation at 15 minutes after tubation | 15 minutes after tubation
  Arterial oxygen saturation (SaO2,%)
Arterial blood hemoglobin at 15 minutes after tubation | 15 minutes after tubation
  Arterial blood hemoglobin (Hb,g/L)
Arterial blood lactate at 15 minutes after tubation | 15 minutes after tubation
  Arterial blood lactate (Lac,mmol/L)
Partial pressure central venous oxygen at 15 minutes after tubation | 15 minutes after tubation
  Partial pressure central venous oxygen(PvO2,mmHg)
Central venous blood oxygen saturation at 15 minutes after tubation | 15 minutes after tubation
  Central venous blood oxygen saturation(ScvO2,%)
Oxygen supply index at 15 minutes after tubation | 15 minutes after tubation
  Oxygen supply index (DO2I,ml/min/m^2)
Calculated index at 15 minutes after tubation | 15 minutes after tubation
  Oxygen consumption index (VO2I,ml/min/m^2)
Partial pressure of oxygen at 30 minutes after tubation | 30 minutes after tubation
  Partial pressure of oxygen (PaO2,mmHg)
Arterial oxygen saturation at 30 minutes after tubation | 30 minutes after tubation
  Arterial oxygen saturation (SaO2,%)
Arterial blood hemoglobin at 30 minutes after tubation | 30 minutes after tubation
  Arterial blood hemoglobin (Hb,g/L)
Arterial blood lactate at 30 minutes after tubation | 30 minutes after tubation
  Arterial blood lactate (Lac,mmol/L)
Partial pressure central venous oxygen at 30 minutes after tubation | 30 minutes after tubation
  Partial pressure central venous oxygen(PvO2,mmHg)
Central venous blood oxygen saturation at 30 minutes after tubation | 30 minutes after tubation
  Central venous blood oxygen saturation(ScvO2,%)
Oxygen supply index at 30 minutes after tubation | 30 minutes after tubation
  Oxygen supply index (DO2I,ml/min/m^2)
Oxygen consumption index at 30 minutes after tubation | 30 minutes after tubation
  Oxygen consumption index (VO2I,ml/min/m^2)
Partial pressure of oxygen at 45 minutes after tubation | 45 minutes after tubation
  Partial pressure of oxygen (PaO2,mmHg)
Arterial oxygen saturation at 45 minutes after tubation | 45 minutes after tubation
  Arterial oxygen saturation (SaO2,%)
Arterial blood hemoglobin at 45 minutes after tubation | 45 minutes after tubation
  Arterial blood hemoglobin (Hb,g/L)
Partial pressure central venous oxygen at 45 minutes after tubation | 45 minutes after tubation
  Partial pressure central venous oxygen(PvO2,mmHg)
Arterial blood lactate at 45 minutes after tubation | 45 minutes after tubation
  Arterial blood lactate (Lac,mmol/L)
Oxygen supply index at 45 minutes after tubation | 45 minutes after tubation
  Oxygen supply index (DO2I,ml/min/m^2)
Oxygen consumption index at 45 minutes after tubation | 45 minutes after tubation
  Oxygen consumption index (VO2I,ml/min/m^2)
Central venous blood oxygen saturation at 45 minutes after tubation | 45 minutes after tubation
  Central venous blood oxygen saturation(ScvO2,%)
Partial pressure of oxygen at the end of surgery | at the end of surgery
  Partial pressure of oxygen (PaO2,mmHg)
Arterial oxygen saturation at the end of surgery | at the end of surgery
  Arterial oxygen saturation (SaO2,%)
Arterial blood hemoglobin at the end of surgery | at the end of surgery
  Arterial blood hemoglobin (Hb,g/L)
Arterial blood lactate at the end of surgery | at the end of surgery
  Arterial blood lactate (Lac,mmol/L)
Partial pressure central venous oxygen at the end of surgery | at the end of surgery
  Partial pressure central venous oxygen(PvO2,mmHg)
Central venous blood oxygen saturation at the end of surgery | at the end of surgery
  Central venous blood oxygen saturation(ScvO2,%)
Oxygen supply index at the end of surgery | at the end of surgery
  Oxygen supply index (DO2I,ml/min/m^2)
Oxygen consumption index at the end of surgery | at the end of surgery
  Oxygen consumption index (VO2I,ml/min/m^2)
Partial pressure of oxygen at 1 minute after extubation | 1 minute after extubation
  Partial pressure of oxygen (PaO2,mmHg)
Arterial oxygen saturation at 1 minute after extubation | 1 minute after extubation
  Arterial oxygen saturation (SaO2,%)
Arterial blood hemoglobin at 1 minute after extubation | 1 minute after extubation
  Arterial blood hemoglobin (Hb,g/L)
Arterial blood lactate at 1 minute after extubation | 1 minute after extubation
  Arterial blood lactate (Lac,mmol/L)
Partial pressure central venous oxygen at 1 minute after extubation | 1 minute after extubation
  Partial pressure central venous oxygen(PvO2,mmHg)
Central venous blood oxygen saturation at 1 minute after extubation | 1 minute after extubation
  Central venous blood oxygen saturation(ScvO2,%)
Oxygen supply index at 1 minute after extubation | 1 minute after extubation
  Oxygen supply index (DO2I,ml/min/m^2)
Oxygen consumption index at 1 minute after extubation | 1 minute after extubation
  Oxygen consumption index (VO2I,ml/min/m^2)
Plartia pressure of oxygen at 5 minutes after extubation | 5 minutes after extubation
  Plartia pressure of oxygen (PaO2,mmHg)
Arterial oxygen saturation at 5 minutes after extubation | 5 minutes after extubation
  Arterial oxygen saturation (SaO2,%)
Arterial blood hemoglobin at 5 minutes after extubation | 5 minutes after extubation
  Arterial blood hemoglobin (Hb,g/L)
Arterial blood lactate at 5 minutes after extubation | 5 minutes after extubation
  Arterial blood lactate (Lac,mmol/L)
Partial pressure central venous oxygen at 5 minutes after extubation | 5 minutes after extubation
  Partial pressure central venous oxnyge(PvO2,mmHg)
Central venous blood oxygen saturation at 5 minutes after extubation | 5 minutes after extubation
  Central venous blood oxygen saturation(ScvO2,%)
Oxygen supply index at 5 minutes after extubation | 5 minutes after extubation
  Oxygen supply index (DO2I,ml/min/m^2)
Oxygen consumption index at 5 minutes after extubation | 5 minutes after extubation
  Oxygen consumption index (VO2I,ml/min/m^2).
mean artery pressure(MAP) after the participants are taken into the operatin after the participantsg room | during surgery
  MAP(mmHg)
heart rate(HR) after the participants are taken into the operating room | during surgery
  HR(beat per minute)
central venous pressure(CVP) after the participants are taken into the operating room | during surgery
  CVP(mmHg)
variability of stroke volume(SVV) after the participants are taken into the operating room | during surgery
  SVV (%)
mean artery pressure(MAP) after the induction | during surgery
  MAP(mmHg)
heart rate(HR) after the induction | during surgery
  HR(heart rate,beat per minute)
central venous pressure(CVP) after the induction | during surgery
  CVP(mmHg)
variability of stroke volume(SVV) after the induction | during surgery
  SVV (variability of stroke volume,%)
mean artery pressure(MAP) at 5 minutes after tubation | 5 minutes after tubation
  MAP(mmHg)m^2)
heart rate(HR) at 5 minutes after tubation | 5 minutes after tubation
  HR(heart rate,beat per minute),
central venous pressure(CVP) at 5 minutes after tubation | 5 minutes after tubation
  CVP(mmHg)
variability of stroke volume(SVV) at 5 minutes after tubation | 5 minutes after tubation
  SVV (variability of stroke volume,%)
mean artery pressure(MAP) at 10 minutes after tubation | 10 minutes after tubation
  MAP(mmHg)
heart rate(HR) at 10 minutes after tubation | 10 minutes after tubation
  HR(heart rate,beat per minute)
central venous pressure(CVP) at 10 minutes after tubation | 10 minutes after tubation
  CVP(mmHg)
variability of stroke volume(SVV) at 10 minutes after tubation | 10 minutes after tubation
  SVV (variability of stroke volume,%)
mean artery pressure(MAP) at 15 minutes after tubation | 15 minutes after tubation
  MAP(mmHg)
heart rate(HR) at 15 minutes after tubation | 15 minutes after tubation
  HR(heart rate,beat per minute)
central venous pressure(CVP) at 15 minutes after tubation | 15 minutes after tubation
  CVP(mmHg)
variability of stroke volume(SVV) at 15 minutes after tubation | 15 minutes after tubation
  SVV (variability of stroke volume,%)
mean artery pressure(MAP) at 30 minutes after tubation | 30 minutes after tubation
  MAP(mmHg)
heart rate(HR) at 30 minutes after tubation | 30 minutes after tubation
  HR(heart rate,beat per minute)
central venous pressure(CVP) at 30 minutes after tubation | 30 minutes after tubation
  CVP(mmHg)
variability of stroke volume(SVV) at 30 minutes after tubation | 30 minutes after tubation
  SVV (variability of stroke volume,%)
mean artery pressure(MAP) at 45 minutes after tubation | 45 minutes after tubation
  MAP(mmHg)
heart rate(HR) at 45 minutes after tubation | 45 minutes after tubation
  HR(heart rate,beat per minute)
central venous pressure(CVP) at 45 minutes after tubation | 45 minutes after tubation
  CVP(mmHg)
variability of stroke volume(SVV) at 45 minutes after tubation | 45 minutes after tubation
  SVV (variability of stroke volume,%)
mean artery pressure(MAP) at the end of surgery | at the end of surgery
  MAP(mmHg)
central venous pressure(CVP) at the end of surgery | at the end of surgery
  CVP(mmHg)
variability of stroke volume(SVV) at the end of surgery | at the end of surgery
  SVV (variability of stroke volume,%)
heart rate(HR) at the end of surgery | at the end of surgery
  HR(heart rate,beat per minute)
mean artery pressure(MAP) at 1 minute after extubation | 1 minute after extubation
  MAP(mmHg)
heart rate(HR) at 1 minute after extubation | 1 minute after extubation
  HR(heart rate,beat per minute)
variability of stroke volume(SVV) at 1 minute after extubation | 1 minute after extubation
  SVV (variability of stroke volume,%)
central venous pressure(CVP) at 1 minute after extubation | 1 minute after extubation
  CVP(mmHg)
mean artery pressure(MAP) at 5 minutes after extubation | 5 minutes after extubation
  MAP(mmHg)
central venous pressure(CVP) at 5 minutes after extubation | 5 minutes after extubation
  CVP(mmHg)
heart rate(HR) at 5 minutes after extubation | 5 minutes after extubation
  HR(heart rate,beat per minute)
variability of stroke volume(SVV) at 5 minutes after extubation | 5 minutes after extubation
  SVV (variability of stroke volume,%)

OTHER OUTCOMES:
Scores of surgical field quality after the induction | during surgery
  Scores of surgical field quality by Fromme et al. and Boezzart et al.(Score 5 means massive uncontrollable bleeding.Score 4 means heavy but controllable bleeding, significant interference with dissection.Score 3 means moderate bleeding,modest compromise of the surgical field. Score 2 means moderate bleeding,nuisance in regard to the surgical field ,but no actual compromise of the ability to dissect.Score 1 means mild bleeding,but no interference with dissection.Score 0 means minimal bleeding,very dry field).
Scores of surgical field quality at 5 minutes after tubation | 5 minutes after tubation
  Scores of surgical field quality by Fromme et al. and Boezzart et al.(Score 5 means massive uncontrollable bleeding.Score 4 means heavy but controllable bleeding, significant interference with dissection.Score 3 means moderate bleeding,modest compromise of the surgical field. Score 2 means moderate bleeding,nuisance in regard to the surgical field ,but no actual compromise of the ability to dissect.Score 1 means mild bleeding,but no interference with dissection.Score 0 means minimal bleeding,very dry field).
Scores of surgical field quality at 10 minutes after tubation | 10 minutes after tubation
  Scores of surgical field quality by Fromme et al. and Boezzart et al.(Score 5 means massive uncontrollable bleeding.Score 4 means heavy but controllable bleeding, significant interference with dissection.Score 3 means moderate bleeding,modest compromise of the surgical field. Score 2 means moderate bleeding,nuisance in regard to the surgical field ,but no actual compromise of the ability to dissect.Score 1 means mild bleeding,but no interference with dissection.Score 0 means minimal bleeding,very dry field).
Scores of surgical field quality at 15 minutes after tubation | 15 minutes after tubation
  Scores of surgical field quality by Fromme et al. and Boezzart et al.(Score 5 means massive uncontrollable bleeding.Score 4 means heavy but controllable bleeding, significant interference with dissection.Score 3 means moderate bleeding,modest compromise of the surgical field. Score 2 means moderate bleeding,nuisance in regard to the surgical field ,but no actual compromise of the ability to dissect.Score 1 means mild bleeding,but no interference with dissection.Score 0 means minimal bleeding,very dry field).
Scores of surgical field quality at 30 minutes after tubation | 30 minutes after tubation
  Scores of surgical field quality by Fromme et al. and Boezzart et al.(Score 5 means massive uncontrollable bleeding.Score 4 means heavy but controllable bleeding, significant interference with dissection.Score 3 means moderate bleeding,modest compromise of the surgical field. Score 2 means moderate bleeding,nuisance in regard to the surgical field ,but no actual compromise of the ability to dissect.Score 1 means mild bleeding,but no interference with dissection.Score 0 means minimal bleeding,very dry field).
Scores of surgical field quality at 45 minutes after tubation | 45 minutes after tubation
  Scores of surgical field quality by Fromme et al. and Boezzart et al.(Score 5 means massive uncontrollable bleeding.Score 4 means heavy but controllable bleeding, significant interference with dissection.Score 3 means moderate bleeding,modest compromise of the surgical field. Score 2 means moderate bleeding,nuisance in regard to the surgical field ,but no actual compromise of the ability to dissect.Score 1 means mild bleeding,but no interference with dissection.Score 0 means minimal bleeding,very dry field).
Scores of surgical field quality at the end of surgery | at the end of surgery
  Scores of surgical field quality by Fromme et al. and Boezzart et al.(Score 5 means massive uncontrollable bleeding.Score 4 means heavy but controllable bleeding, significant interference with dissection.Score 3 means moderate bleeding,modest compromise of the surgical field. Score 2 means moderate bleeding,nuisance in regard to the surgical field ,but no actual compromise of the ability to dissect.Score 1 means mild bleeding,but no interference with dissection.Score 0 means minimal bleeding,very dry field).
Scores of surgical field quality at 5 minutes after extubation | 5 minutes after extubation
  Scores of surgical field quality by Fromme et al. and Boezzart et al.(Score 5 means massive uncontrollable bleeding.Score 4 means heavy but controllable bleeding, significant interference with dissection.Score 3 means moderate bleeding,modest compromise of the surgical field. Score 2 means moderate bleeding,nuisance in regard to the surgical field ,but no actual compromise of the ability to dissect.Score 1 means mild bleeding,but no interference with dissection.Score 0 means minimal bleeding,very dry field).
Scores of surgical field quality at 1 minute after extubation | 1 minute after extubation
  Scores of surgical field quality by Fromme et al. and Boezzart et al.(Score 5 means massive uncontrollable bleeding.Score 4 means heavy but controllable bleeding, significant interference with dissection.Score 3 means moderate bleeding,modest compromise of the surgical field. Score 2 means moderate bleeding,nuisance in regard to the surgical field ,but no actual compromise of the ability to dissect.Score 1 means mild bleeding,but no interference with dissection.Score 0 means minimal bleeding,very dry field).
operation time after the induction | during surgery
  operation time（minutes）
operation time after the participants are taken into the operating room | during surgery
  operation time（minutes）
operation time at 5 minutes after tubation | 5 minutes after tubation
  operation time（minutes）
operation time at 10 minutes after tubation | 10 minutes after tubation
  operation time（minutes）
operation time at 15 minutes after tubation | 15 minutes after tubation
  operation time（minutes）
operation time at 30 minutes after tubation | 30 minutes after tubation
  operation time（minutes）
operation time at 45 minutes after tubation | 45 minutes after tubation
  operation time（minutes）
operation time at the end of surgery | at the end of surgery
  operation time（minutes）
operation time at 5 minutes after extubation | 5 minutes after extubation
  operation time（minutes）
operation time at 1 minute after extubation | 1 minute after extubation
  operation time（mintes）
estimated blood loss after the induction | during surgery
  estimated blood loss（ml）
estimated blood loss after the participants are taken into the operating room | during surgery
  estimated blood loss（ml）
estimated blood loss at 5 minutes after tubation | 5 minutes after tubation
  estimated blood loss（ml）
estimated blood loss at 10 minutes after tubation | 10 minutes after tubation
  estimated blood loss（ml）
estimated blood loss at 15 minutes after tubation | 15 minutes after tubation
  estimated blood loss（ml）
estimated blood loss at 30 minutes after tubation | 30 minutes after tubation
  estimated blood loss（ml）
estimated blood loss at 45minutes after tubation | 45 minutes after tubation
  estimated blood loss（ml）
estimated blood loss at the end of surgery | at the end of surgery
  estimated blood loss（ml）
estimated blood loss at 1 minute after extubation | 1 minute after extubation
  estimated blood loss（ml）
estimated blood loss at 5 minutes after extubation | 5 minutes after extubation
  estimated blood loss（ml）
Scores of surgical field quality after the participants are taken into the operating room | during surgery
  Scores of surgical field quality by Fromme et al. and Boezzart et al.(Score 5 means massive uncontrollable bleeding.Score 4 means heavy but controllable bleeding, significant interference with dissection.Score 3 means moderate bleeding,modest compromise of the surgical field. Score 2 means moderate bleeding,nuisance in regard to the surgical field ,but no actual compromise of the ability to dissect.Score 1 means mild bleeding,but no interference with dissection.Score 0 means minimal bleeding,very dry field).

CONTACTS AND LOCATIONS:
Overall Officials: Cao Yang, Study Director — Guangzhou Red Cross Hospital
Locations (1):
- Guangzhou Red cross hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kako H, Gable A, Martin D, Beebe A, Thung A, Samora W, Klamar J, Bhalla T, Tobias JD. A prospective, open-label trial of clevidipine for controlled hypotension during posterior spinal fusion. J Pediatr Pharmacol Ther. 2015 Jan-Feb;20(1):54-60. doi: 10.5863/1551-6776-20.1.54. PMID 25859171
- [Background] Amr YM, Amin SM. Effects of preoperative beta-blocker on blood loss and blood transfusion during spinal surgeries with sodium nitroprusside-controlled hypotension. Saudi J Anaesth. 2012 Jul;6(3):263-7. doi: 10.4103/1658-354X.101219. PMID 23162401